CLINICAL TRIAL: NCT03432949
Title: Radium-223 Combined With Dexamethasone as First-line Therapy in Patients With Metastatic Castrate Resistant Prostate Cancer
Brief Title: Radium-223 Combined With Dexamethasone as First-line Therapy in Patients With M+CRPC
Acronym: TRANCE
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Health Network, Toronto (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17-5196
Record Dates: First submitted 2018-01-30; First posted 2018-02-14 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: Metastatic Prostate Cancer
Keywords: Radium-223; Dexamethasone; mCRPC
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Dexamethasone; Radium-223; Calcium Dobesilate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard of Care Radium-223 (No Intervention): Radium-223 treatment will be administered as per standard of care.
- Radium-223 with oral Dexamethasone 0.5 mg (Experimental): Dexamethasone will be administered as 0.5 mg capsules by mouth per day during the duration of the Radium-223 treatment.
  Interventions: Drug: Dexamethasone plus Radium-223

INTERVENTIONS:
Drug: Dexamethasone plus Radium-223 — Dexamethasone will be administered as 0.5 mg capsules by mouth per day during the duration of the Radium-223 treatment.
  Other Names: Dexamethasone; Baycadron
  Arms: Radium-223 with oral Dexamethasone 0.5 mg

SUMMARY:
More than 90% of patients with metastatic castration-resistant prostate cancer (mCRPC) no longer responding to androgen deprivation hormonal therapy have evidence of bone metastases. This is a major cause of death, disability, and decreased quality of life.

Radium-223 is radiopharmaceutical meaning that the drug is a radioactive compound used for therapeutic purposes. It is given intravenously (through a vein) every 4 weeks for 6 cycles. Research has demonstrated safety and efficacy in mCRPC patients resulting in radium-223 becoming a standard of care option for such patients in addition to chemotherapy and new oral hormonal drugs enzalutamide or abiraterone.

Prior research studies using radium-223 have shown improved survival in about 30% of patients. The same studies in combination with data collected from clinical use have also shown that between 20 and 50% of men do not complete the full 6 cycle course of treatment due to side effects or a rise in prostate specific antigen (PSA) requiring the stoppage of radium-223 therapy to start one of the other drug therapies.

The purpose of this study is to determine whether an oral drug called dexamethasone (a corticosteroid) given together with radium-223 may control PSA levels and reduce side effects during radium-223 treatment. Corticosteroids are anti-inflammatory medicines prescribed for a broad range of conditions and are widely used in conjunction with chemotherapy treatments for cancer. Prior research studies have shown that dexamethasone reduces PSA levels by lowering the production of androgens (i.e. male hormones) and improves overall tolerance for cancer-fighting drugs and therapies.

Up to 24 men being treated with radium-223 at University Health Network will be enrolled into this study. If the study is positive, it might offer an improved quality of life and extended survival.

ELIGIBILITY:
INCLUSION CRITERIA:

1. Clinical diagnosis of prostate cancer
2. ECOG status ≤ 2
3. PSA ≥ 2.0 ng/mL
4. Rising PSA in combination with new metastases or evidence of radiographic disease progression despite castrate levels of testosterone while on androgen deprivation therapy (ADT) or following bilateral orchiectomy
5. Symptomatic disease defined as any analgesic use for pain or receipt of radiotherapy for bony metastatic disease
6. Adequate renal and hepatic function:

   * Cr ≤ 1.5 x upper limit of normal (ULN)
   * AST ≤ 2.5 x ULN
   * ALT ≤ 2.5 x ULN
   * Albumin > 25 g/L
   * Total bilirubin ≤ 1.5 x ULN
7. Adequate hematologic function

   * Absolute neutrophil count (ANC) ≥ 1.5 x 109/L
   * Platelet count ≥ 100 x 109/L
   * Hemoglobin ≥ 100 g/L
8. Evidence of bone metastasis on bone scan, CT, MRI or PET
9. Life expectancy ≥ 6 months

EXCLUSION CRITERIA:

1. Visceral metastatic PCa (brain, liver, lung, bulky adenopathy). Note that metastatic lymphadenopathy < 3cm is acceptable for inclusion as long as there is evidence of bone metastasis.
2. Previous treatment with abiraterone, enzalutamide, docetaxel or other systemic chemotherapy for PCa
3. Imminent spinal cord compression or history of spinal cord compression
4. Previous treatment with systemic corticosteroids for PCa at any time
5. Contraindication to receipt of systemic corticosteroids (i.e. uncontrolled diabetes)
6. Prior or current enrolment in any other interventional clinical trial

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2018-02-23 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2024-07-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of total doses delivered on schedule | Through infusion completion, an average of 24 weeks
  To assess the feasibility of delivering 6-treatment cycles of Radium-223 without delays when administered in combination with low-dose oral dexamethasone for patients with metastatic CRPC and bony metastases who are abiraterone, enzalutamide and systemic chemotherapy naïve.

CONTACTS AND LOCATIONS:
Locations (1):
- University Health Network, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No